CLINICAL TRIAL: NCT03847220
Title: Prospective Study of the Utility of the BOMET-QOL Questionnaire Patients With Breast Cancer and Bone Metastasis
Brief Title: Study of the Utility of the BOMET-QOL Questionnaire Patients With Breast Cancer and Bone Metastasis
Acronym: MAbomet
Status: Completed | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Mabomet
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Carcinoma Metastatic to the Bone
Keywords: metastatic breast cancer; bone metastasis; quality of life; psychometric; treatment; assessments
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BOMET-QoL questionnaire — study to evaluate the utility of the BOMET-QoL questionnaire in patients with BC and BM

SUMMARY:
Epidemiological, prospective and multicenter study to evaluate the utility of the BOMET-QoL questionnaire in patients with breast cancer (BC) and bone metastases (BM).

DETAILED DESCRIPTION:
Population: Patients over 18 with breast cancer and bone metastasis.

Inclusion criteria:

* Patient over 18 years of age.
* Patient diagnosed with breast cancer (BC) and bone metastases (BM).
* Patient who has granted informed consent in writing to participate in the study.
* Patient capable of understanding and completing the questionnaires.

Exclusion criteria:

* Patient with another type of disease that, in the investigator's opinion, could mask the study results.
* Patients with a life expectancy of less than 8 months.
* Patient who is participating in a clinical trial with an unregistered drug at the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age.
* Patient diagnosed with BC and BM.
* Patient who has granted informed consent in writing to participate in the study.
* Patient capable of understanding and completing the questionnaires

Exclusion Criteria:

* Patient with another type of disease that, in the investigator's opinion, could mask the study results.
* Patients with a life expectancy of less than 8 months.
* Patient who is participating in a clinical trial with an unregistered drug at the start of the study.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — female patient over 18 years of age
Study Population: The patients susceptible for inclusion in the study were women with breast cancer and bone metastasis in any location who met the screening criteria described in the study protoco
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2007-10-23 (Actual); Primary Completion 2010-05-20 (Actual); Study Completion 2012-07-07 (Actual)

PRIMARY OUTCOMES:
Impact on the HRQoL | Up to 24 months
  Impact on the HRQoL of patients with BC and BM will be measured by the BOMET-QoL questionnaire in the context of normal clinical practice. The questionnaire will be administered to patients in each study visit from baseline visit to the final visit at 24 months. The score of the questionnaire will be measured as: Score: 0 - Always, 1 - Nearly always, 2 - Sometimes, 3 - Rarely, 4 - Never, were never is the best option and always means patient has a bad health condition.

SECONDARY OUTCOMES:
Measurement properties of the BOMET-QoL questionnaire: validity | Up to 24 months
  Its cross-sectional validity will be evaluated by analysing the relationship between the BOMET-QoL scores and different clinical variables (presence of Skeleton-Related Event (SREs), symptoms and Eastern Cooperative Oncology Group (ECOG) index). The relationship between the pain VAS score and the question about state of health perceived by patient with HRQoL according to BOMET-QoL will be analysed.
Measurement properties of the BOMET-QoL questionnaire: feasibility | Up to 24 months
  BOMET-QoL will be considered rapidly completed if patients complete questionnaire in less than 10 minutes.
Measurement properties of the BOMET-QoL questionnaire: sensitivity to change | Up to 24 months
  Sensitivity to change can be evaluated by calculating the effect size or the Minimum Clinically Important Difference, as statistics based on effect size provide direct information about the magnitude of the change, expressed as a variation, also used to calculate the Minimum Clinically Important Difference.
Impact of skeletal-related events (SREs) on HRQoL (BOMET-QoL scores) | Up to 24 months
  The impact of skeletal-related events (SREs) on HRQoL (BOMET-QoL scores) will be measured by comparing patients who presented SREs with patients with without SREs.
Relation between Eastern Cooperative Oncology Group (ECOG) and HRQoL (BOMET-QoL scores). | Up to 24 months
  ECOG: This scale consists of 5 levels (0 = No restrictions to carry out the activities normal, 1 = Restrictions to perform vigorous physical activities. It has the capacity to perform ambulation and light work, 2 = Ability to ambulate and perform personal care but not able to work. Capacity for standing and walking for> 50% of waking hours, 3 = Able to perform care limited personal; Incarcerated or restrained to be in a chair for> 50% of the hours of vigil, 4 = complete disability; he can not perform any personal care; it remains in bed or in a chair all the time, 5 = Death). In it the observer assesses the state of symptoms and the level of functioning in relation to ambulatory status and need for care. Patients with an Eastern Cooperative Oncology Group (ECOG) functional scale between 0-1 will obtain a higher score (better HRQoL) in the BOMET-QoL questionnaire.
Correlation between visual analogue scale (VAS) score of pain and HRQoL (BOMET-QoL scores). | Up to 24 months
  At the baseline visit, patients who obtain higher scores on the Analogue Visual Pain Scale will obtain a lower score (worse HRQOL) in the BOMET-QoL questionnaire. Correlation between the BOMET-QoL scores and the pain VAS scores regarding whether it improves, stays the same or gets worse between the different study visits. VAS: 0 no pain - 10 unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (15):
- Spain (15):
  - Hospital Universitario Virgen Del Rocío, Seville, Andalusia
  - Hospital General de Guadalajara, Guadalajara, Castille-La Mancha
  - ICO Badalona Hospital Universitari Germans Trias I Pujol, Badalona, Catalonia
  - Hospital Universitari Clinic I Provincial, Barcelona, Catalonia
  - Hospital Santa Creu I Sant Pau, Barcelona, Catalonia
  - Hospital Mutua de Terrassa, Barcelona, Catalonia
  - ICO Girona Hospital Dr. Josep Trueta, Girona, Catalonia
  - Hospital Universitari Arnau de Vilanova, Lleida, Catalonia
  - Fundació Althaia, Xarxa Assistencial de Manresa, Manresa, Catalonia
  - Hospital General Universitario de Alicante, Alicante, Cominidad Valenciana
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Centro Oncologico de Galicia, A Coruña, Galicia
  - Complejo Hospitalario de Pontevedra, Pontevedra, Galicia
  - Hospital de Barbastro, Barbastro, Huesca
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Barnadas A, Munoz M, Margeli M, Chacon JI, Cassinello J, Antolin S, Adrover E, Ramos M, Carrasco E, Jimeno MA, Ojeda B, Gonzalez X, Gonzalez S, Constenla M, Florian J, Miguel A, Llombart A, Lluch A, Ruiz-Borrego M, Colomer R, Del Barco S; GEICAM, Spanish Breast Cancer Group. BOMET-QoL-10 questionnaire for breast cancer patients with bone metastasis: the prospective MABOMET GEICAM study. J Patient Rep Outcomes. 2019 Dec 21;3(1):72. doi: 10.1186/s41687-019-0161-y. PMID 31865481
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org